CLINICAL TRIAL: NCT00838643
Title: Incidence of Invasive Aspergillosis in Allogeneic Stem Cell Transplantation Patients: an Italian Prospective Multicentre Study
Brief Title: Invasive Aspergillosis After Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ospedale Santa Croce-Carle Cuneo (Other)
Responsible Party: Nicola Mordini, Ospedale Santa Croce-Carle Cuneo
Other Study IDs: Gal-01
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Hematological Diseases; Invasive Aspergillosis
Keywords: allogeneic transplantation; Invasive aspergillosis
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Allogeneic pts: Adult allogeneic HSCT recipients

SUMMARY:
Evaluation of incidence of invasive aspergillosis in patients who have undergone an allogeneic stem cell transplantation, with particular regard to the role of galactomannan assay and of early TC scan in asymptomatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 16 years
* Allogeneic HSCT for a haematological disease
* Written informed consent to the study

Exclusion Criteria:

* Pediatric patients

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients given allogeneic HSCT in tertiary care centers or university hospitals in Piedmont
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2002-05; Primary Completion 2007-06 (Actual); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of invasive aspergillosis | 1 year

SECONDARY OUTCOMES:
Clinical applicability of the EORTC/MSG criteria in a prospective multicenter trial | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Sanitaria Ospedaliera santa Croce e Carle, Cuneo, Italy